CLINICAL TRIAL: NCT03802994
Title: Immune Response to Pneumococcal Vaccination in Aging Renal Transplant Recipients
Brief Title: Pneumococcal Conjugate Vaccine in Aging Renal Transplant
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Due to COVID pandemic further recruitment of subjects was unethical.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INFB-019-17F; CX001568 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2018-12-18; First posted 2019-01-14 (Actual); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Renal Transplantation; Aging
Keywords: Prevnar; pneumococcal conjugate vaccine; aging; renal transplant recipient
MeSH Terms: interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Immune response to immunization with Prevnar in elderly aging renal transplant compared to comparison groups: healthy young, healthy elderly, healthy elderly hypertension (HTN) and young renal transplants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- 1.Aging RT (Experimental): Renal transplant recipients between 65-75 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause or renal failure was either DMII or HTN.
  Interventions: Other: Peripheral blood sample
- 2.Young RT (Active Comparator): Renal transplant recipients between 35-45 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause or renal failure was either DMII or HTN.
  Interventions: Other: Peripheral blood sample
- 3.Healthy elderly (Active Comparator): Healthy persons between the ages 65-75 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  Interventions: Other: Peripheral blood sample
- 4.Elderly DMII or HTN and normal renal function (Active Comparator): Persons between the ages 65-75 with DMII or hypertension but normal renal function who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  Interventions: Other: Peripheral blood sample
- 5.Healthy young (Experimental): Healthy persons between the ages 35-45 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23) or are willing to receive PPV23 and 1 year later Prevnar 13.
  Interventions: Drug: 23 valent pneumococcal polysaccharide vaccine; Biological: 13 valent conjugated pneumococcal vaccine; Other: Peripheral blood sample

INTERVENTIONS:
Drug: 23 valent pneumococcal polysaccharide vaccine — FDA approved pneumococcal polysaccharide vaccine containing capsular polysaccharide of 23 different pneumococcal serotypes. Only group 5 will potentially receive this as an intervention.
  Other Names: Pneumovax 23 or PPV23
  Arms: 5.Healthy young
Biological: 13 valent conjugated pneumococcal vaccine — FDA approved pneumococcal polysaccharide vaccine containing capsular polysaccharide of 13 different pneumococcal serotypes conjugated to CRM197. Only group 5 will receive this as an intervention. In all other groups Prevnar 13 will be given as standard of care.
  Other Names: Prevnar 23 or PCV13
  Arms: 5.Healthy young
Other: Peripheral blood sample — Peripheral blood samples (30-60 mL) will be collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) for groups 1-4 and at days 366, 373 and 396 for group 5. In addition, day 5, and 10 blood samples will be obtained from a limited (n=10) number of elderly RT participants to determine the optimal time point for circulation of PPS-specific B cells. Yearly blood samples will be obtained thereafter for serum antibody and OPA analyses to test longevity of antibody and OPA responses. Samples obtained from days 0, 30 and yearly samples will be used for antibody titers and opsonophagocytic assays. Samples from day 0 (day of vaccination with PCV13) and day 7 will be used for flow cytometric analysis.
  Other Names: blood draw

SUMMARY:
The goal of the research proposed in the current application is to first define how much antibody aging renal transplant and dialysis recipients make after they are vaccinated with the pneumonia vaccine and how this compares to similar aged persons with good renal function and healthy young adults. The investigators will study differences in the kind of B cells and markers on the B cells that are known to be important in the response to the pneumonia vaccine in aging renal transplant and aging dialysis recipients compared to similarly aged and young healthy controls. Finally, the investigators will study how safe the pneumonia vaccine is in aging renal transplants. The answers to these questions will help in designing a better vaccine for older people with a renal transplant or on dialysis.

DETAILED DESCRIPTION:
Objectives / Specific Aims

Individuals >65 years of age, are the most rapidly growing population amongst those with end stage renal disease (ESRD) and account for more than 18% of renal transplant (RT) recipients.

The incidence of pneumococcal disease is significantly higher in both elderly and those with RT and the combination of these factors is likely additive, if not synergistic, for invasive pneumococcal disease (IPD). It is recommended that both elderly>65 and RT recipients be vaccinated with a regimen that includes both the 13-valent pneumococcal conjugate vaccine (PCV13) and the 23-valent pneumococcal polysaccharide vaccine (PPV23). However, small immunogenicity studies performed in the transplant populations have not shown superiority of a PCV containing regimen. Moreover, the addition of PCV to the pneumococcal vaccine regimen does not improve protective immunity in this population. Studies to date fail to elucidate the possible foundation of the disappointing immune responses to the PCV regimens.

Specific Aim 1. The investigators will define immune responses by measuring serum antibody and functional antibody responses to PPS 14, 19A and 23F following PCV13 vaccination in RT recipients 65-75 years of age and compare these to: RT recipients 35-45 years of age and persons with DM/HTN but normal function 65-75 years of age to dissect out the age and RT components respectively. Healthy persons 35-45 and 65-75 years of age will be studied as age appropriate reference.

Specific Aim 2. The investigators will measure and characterize the antigen-specific B cell subset response following immunization with PCV13 in the RT recipients 65-75 years of age and compare them to each of the groups described in Specific Aim 1 using flow cytometry and fluorescently labeled PPS and monoclonal antibodies. These measures will be correlated with post-immunization functional antibody activity, a surrogate of protection.

Specific Aim 3. The investigators will measure TNFR expression by B cells following immunization with PCV13 in 65-75 year old RT and compare them to each of the groups described in Specific Aim 1. Gene expression, with focus on the B cell activating factor (BAFF) system, will be measured in PPS-specific and non-PPS specific B cells using single cell genomics and flow cytometry. These measures will be correlated with post-immunization functional antibody activity, a surrogate of protection.

The central hypothesis is that the aging RT population responds poorly to PCV13 vaccination reflecting the combined effects of aging and RT. The investigators postulate that both the number of memory B cells and expression of tumor necrosis factor (TNF) superfamily receptors, which play crucial roles in the response to pneumococcal polysaccharides (PPS), are deficient in the elderly RT population and contribute to poor pneumococcal vaccine responses.

The investigators have developed fluorescently labeled PPS allowing us to study the nature and surface receptors of PPS-specific B cells. The preliminary data demonstrate that RT recipients 1. Respond poorly to pneumococcal immunization as measured by antibody titer and functional antibody activity. 2. RT recipients and healthy elderly have lower absolute number of both IgM and switched memory B cells. 3. The number of PPS-specific IgM and switched memory B cells are significantly lower in RT recipients and 4. TACI and BAFF-R, members of the TNF superfamily receptors, expression is significantly lower in the PPS-specific memory B cells in the RT population versus healthy controls. The overall objective of this proposal is to characterize the immune response and explore possible mechanisms of poor vaccine responsiveness following immunization with PCV in the rapidly growing group of elderly with RT. As the RT population is a heterogeneous group the investigators will study only those in whom the underlying cause of renal failure is diabetes mellitus type 2 (DM2) and/or hypertension (HTN).

Intervention to be studied The intervention to be studied is the immune response to immunization with PCV13 or Prevnar13. This FDA approved vaccine is given as part of the standard of care in Groups 1-4. The experimental part of the protocol in these groups will be blood draws at days 0, 7, 30 and years 1 and 2 in these groups.

In Group 5 two interventions will occur: 1. Immunization with the FDA approved PPV23 or Pneumovax 23 and 2. PCV13 a FDA approved vaccine. In addition, blood samples will be obtained at days 0, 7, 30 year 1 and year2.

Both PPV23 and PCV13 are FDA approved vaccines for use in humans. PCV13 is recommended for all individuals enrolled in Groups 1-4. It is not recommended as routine part of care in Group 5 enrolled individuals however it has never shown to be harmful in this group of individuals.

Study Endpoints The primary endpoint of this study is: quantify the antibody titers in mg/mL and opsonophagocytic antibody titer calculated as serum dilution, number of polysaccharide specific B cells, and absolute number of cells/mL induced by vaccination with PCV13.

Secondary endpoint of the study is to describe differences in gene expression of 56 genes to be determined by single cell PCR and comparing these between groups.

The primary safety endpoint of the study is measured as minimal versus moderate local side effect. Minimal side effect measured as no impairment in activity. Moderate local side effect is a side effect affecting use of the extremity for less than 24 hours.

Inclusion and Exclusion Criteria/ Study Population: as described in inclusion/exclusion section

Diversity: the investigators will attempt to mimic the local renal transplant recipient population consisting of a disproportionately high number of males (>60%) of African-American decent, 50%.

Number of Subjects 275

Study Sites

1. The MUSC Renal Transplant clinic is located on the 9th floor of the Rutledge Tower
2. The nephrology clinic at the Ralph H. Johnson VA Medical Center
3. the P.I.'s laboratory at the Strom Thurmond Building Room 411

Recruitment Methods

* Potential study participants will be recruited from Ralph H. Johnson Veterans Affair Medical Center and Medical University of South Carolina during the appointment with their treating physician. Flyers will be posted in the waiting room areas of the clinics and attending physicians and clinic nurses will be asked to keep this study in mind and mention availability of these studies to their patients when ordering PCV13 for them.
* Potential study subjects will be identified by reviewing medical records and by physician's recommendations.
* Flyers will be used to recruit study subjects as well as broadcast emails for MUSC and VA employees and volunteers.

Consent Process

Informed Consent will be obtained in a private room from all participants at either:

1. The MUSC Renal Transplant clinic is located on the 9th floor of the Rutledge Tower Or 2.The nephrology clinic at the Ralph H. Johnson VA Medical Center Or 3. the P.I.'s laboratory at the Strom Thurmond Building Room 411

Consent will be sought of competent adults who express interest in the study. The purpose of the study, the study details regarding gathering health information and obtaining blood samples, the potential benefit and risks involved, including risk of blood draw and vaccination, will be explained in detail and in layman terms, as well as the non-standard of care explained to the potential subject (i.e. blood draws for groups 1-4, vaccination protocol and blood draws for group 5).

Study Design / Methods The overall objective of this proposal is to characterize the immune response and explore possible mechanisms of poor vaccine responsiveness following immunization with PCV in the rapidly growing group of elderly with RT. As the RT population is a heterogeneous group the investigators will study only those in whom the underlying cause of renal failure is diabetes mellitus type 2 (DM2) and/or hypertension (HTN). There will be 5 study groups as outlined above.

results obtained in various groups will be compared.

Timing of blood samples Peripheral blood samples will be collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) for groups 1-4 and at days 366, 373 and 396 for group 5. BAFF concentration will be measured at day

The vaccine(s) administered to the participants are FDA approved vaccinations and vaccination protocols. The standard and recommended dose of vaccine will be administered either by a qualified nurse or physician and both vaccines are considered low risk. In groups 1-4 PCV13 will be administered per standard of care and is not part of the experimental protocol. In group 5, both PPV23 and PCV 13 are not routine part of care and are part of the experimental protocol. These vaccines have however been extensively studied in this and other populations and are considered low risk and 70-80% protective against pneumococcal disease.

The risk associated with blood draws is minimal.

* Pre- and post-immunization serum antibody titers and opsonophagocytic antibody titers to PPS14, 19A and 23F in ug/mL determined by ELISA IgM and switched memory B cell number and percentage determined by flow cytometry
* PPS+ B cell number and percentage determined by flow cytometry
* Serum BAFF concentration by ELISA
* Gene expression of 56 genes will be studies using single cell PCR analysis

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are group specific. HBV, HCV and HIV testing are not necessary in the RT groups as all RT recipients are tested prior to transplant. The investigators will not restrict volunteers with respect to gender, ethnic or racial group.

Groups 1 (65-75 yrs) and 2 (35-45 yrs) Renal Transplant populations

* End stage renal disease cause either DM2 and/or hypertension (HTN)
* Renal transplant >12 months ago

Group 3: Diabetic/hypertensive 65-75 year old controls

* With DM2 and/or HTN
* Previous immunization with PPV23 >1 year prior
* Willingness to be tested for HIV, HBV and HCV
* "normal kidney function" defined as glomerular filtration rate (GFR) of 60% or above

Group 4: Healthy Control 65-75 yr old

* Without DM2
* May have high blood pressure (systolic>140 and/or diastolic>90) as long as it is well controlled (systolic<140 and/or diastolic <90) and has not affected kidney function.
* Previous receipt of PPV23 > 1 year prior
* Willingness to be tested for HIV, HBV and HCV

Group 5: Healthy Control 35-45 yr old

* Without DM2.
* May have high blood pressure (systolic>140 and/or diastolic>90) as long as it is well controlled (systolic<140 and/or diastolic <90) and has not affected kidney function.
* Willingness to be tested for HIV, HBV and HCV and filling out a medical questionnaire that will include diabetes screening.

Exclusion Criteria:

Exclusion criteria are either applicable to all groups or group specific. Therefore we have listed the exclusion criteria applicable to ALL groups first. Group specific criteria are listed under each group.

Exclusion Criteria common to all groups

* Previous immunization with PCV13.
* Pregnancy, no contraceptive practice in women of childbearing age, or breastfeeding
* Known anaphylaxis, hypersensitivity or "bad allergic reaction" to the pneumonia vaccine. This does not include egg allergy or previous Guillan Barre syndrome.
* Those who received blood products or gamma globulin within 3 months.
* Inability to comprehend or sign the informed consent form
* Previous/present illness that may affect immune response to the vaccine

  * previous pneumococcal disease
  * disease
  * removal of the spleen
  * auto-immune disease such as lupus or rheumatoid arthritis
  * end-stage liver disease
  * cancer
* Significant abnormalities (3xULN and all those considered to be critical values) in CBC, chemistries including glucose.
* HIV, HBsAg or HCV positivity
* Receipt of PPV23 within 1 year

Groups 1 (65-75 yrs) and 2 (35-45 yrs) Renal Transplant populations

* Medications that are known to affect immune function (chemotherapy, anti-TNF agents) with the exception of anti-rejection medication.
* Episode of acute rejection within the last 6 month period

Group 3: Diabetic/hypertensive 65-75 year old controls

* Medications that are known to affect immune function (chemotherapy, anti-TNF agents).
* The inclusion/exclusion criteria will be determined by chart review.

Group 4: Healthy Control 65-75 yr old

* Medications that are known to affect immune function (chemotherapy, anti-TNF agents).
* The inclusion/exclusion criteria will be determined by chart review and pregnancy test for females of child bearing potential.

Group 5: Healthy Control 35-45 yr old

* Medications that are known to affect immune function (chemotherapy, anti-TNF agents).
* The inclusion/exclusion criteria will be determined by chart review and pregnancy test for females of child bearing potential.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Westerink, MD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (2):
- United States (2):
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: prevnar vaccine
Period: Overall Study
Arm/Group | 1.Aging RT | 2.Young RT | 3.Healthy Elderly | 4.Elderly DMII or HTN and Normal Renal Function | 5.Healthy Young
Started | 9; 9 prevnar vaccine | 12; 12 prevnar vaccine | 15; 15 prevnar vaccine | 11; 11 prevnar vaccine | 10; 10 prevnar vaccine
Completed | 9; 9 prevnar vaccine | 10; 10 prevnar vaccine | 12; 12 prevnar vaccine | 9; 9 prevnar vaccine | 8; 8 prevnar vaccine
Not Completed | 0; 0 prevnar vaccine | 2; 2 prevnar vaccine | 3; 3 prevnar vaccine | 2; 2 prevnar vaccine | 2; 2 prevnar vaccine
Not completed — Lost to Follow-up | 0 | 2 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Population: In Groups 1, 3,4 and 5 2 individuals per group were enrolled but did not complete the study which affected parameters of all study objectives: pre- to post-antibody and opsonophagocytic responses, B cell analysis and inflammatory markers.
Groups:
- 1.Aging RT: Renal transplant recipients between 65-75 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause or renal failure was either DMII or HTN.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples obtained from days 0 and 30 were used for antibody titers and opsonophagocytic assays. Samples from day 7 was used for flow cytometric analysis.
- 2.Young RT: Renal transplant recipients between 35-45 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause or renal failure was either DMII or HTN.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples obtained from days 0, 30 were used for antibody titers and opsonophagocytic assays. Samples from day 7 were used for flow cytometric analysis.
- 3.Healthy Elderly: Healthy persons between the ages 65-75 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23). Samples obtained from days 0, 30 were used for antibody titers and opsonophagocytic assays. Samples from day 7 was used for flow cytometric analysis.
- 4.Elderly DMII or HTN and Normal Renal Function: Persons between the ages 65-75 with DMII or hypertension but normal renal function who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30. Samples from day 7 were used for flow cytometric analysis.
- 5.Healthy Young: Healthy persons between the ages 35-45 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23).
  23 valent pneumococcal polysaccharide vaccine: FDA approved pneumococcal polysaccharide vaccine containing capsular polysaccharide of 23 different pneumococcal serotypes. All young healthy participants recruited were already immunized with pneumovax at least one year prior to enrollment
  13 valent conjugated pneumococcal vaccine: FDA approved pneumococcal polysaccharide vaccine containing capsular polysaccharide of 13 different pneumococcal serotypes conjugated to CRM197 was adminstered at day 0. Only group 5 received this as an intervention. In all other groups Prevnar 13 was given as standard of care.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples obtained from days 0, 30 were used for antibody titers and opsonophagocytic assays. Samples from day 7 were used for flow cytometric analysis.
- Total: Total of all reporting groups
Arm/Group | 1.Aging RT | 2.Young RT | 3.Healthy Elderly | 4.Elderly DMII or HTN and Normal Renal Function | 5.Healthy Young | Total
Number analyzed (Participants) | 9 | 12 | 15 | 11 | 10 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 12 | 0 | 0 | 10 | 22
  >=65 years | 9 | 0 | 15 | 11 | 0 | 35
Age, Continuous [Median (Full Range); unit: years] | 67 [65 to 71] | 41 [35 to 45] | 66 [65 to 69] | 66 [65 to 72] | 40 [35 to 44] | 65 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 0 | 0 | 2 | 7
  Male | 8 | 8 | 15 | 11 | 8 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 9 | 9 | 6 | 2 | 35
  White | 0 | 3 | 6 | 5 | 8 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 12 | 15 | 11 | 10 | 57

OUTCOME MEASURES:

1. Primary Outcome: Anti-pneumococcal IgG Antibody (ug/ml) Change
Description: Measure the opsonic antibody response against streptococcus pneumonia serotypes 14, 19A and 23F at days 0 and 30.
  Comparing elderly RT recipients versus healthy elderly and elderly with DM/HTN.
Time Frame: Baseline, 30 days
Population: Participants who completed PCV13 immunization and from whom blood samples were obtained on day 0, 7, and 30.
  There is thus a discrepancy between the number of enrolled and analyzed participants in groups 2,3,4 and 5.
Measure: Geometric Mean (Standard Deviation); unit: microgram/ml
Groups:
- 1.Aging RT: Renal transplant recipients between 65-75 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause or renal failure was either DMII or HTN.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples obtained from days 0 and 30 were used for antibody titers and opsonophagocytic assays. Samples from day 7 were used for flow cytometric analysis.
- 2.Young RT: Renal transplant recipients between 35-45 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause or renal failure was either DMII or HTN.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples obtained from days 0 and 30 were used for antibody titers and opsonophagocytic assays. Samples from day 7 were used for flow cytometric analysis.
- 3.Healthy Elderly: Healthy persons between the ages 65-75 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples obtained from days 0 and 30 were used for antibody titers and opsonophagocytic assays. Samples from day 7 were used for flow cytometric analysis.
- 4.Elderly DMII or HTN and Normal Renal Function: Persons between the ages 65-75 with DMII or hypertension but normal renal function who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples obtained from days 0 and 30 were used for antibody titers and opsonophagocytic assays. Samples from day 7 were used for flow cytometric analysis.
- 5.Healthy Young: Healthy persons between the ages 35-45 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  13 valent conjugated pneumococcal vaccine: FDA approved pneumococcal polysaccharide vaccine containing capsular polysaccharide of 13 different pneumococcal serotypes conjugated to CRM197 was used for immunization at day 0. Only group 5 received this as an intervention. In all other groups Prevnar 13 will be given as standard of care.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples obtained from days 0 and 30 were used for antibody titers and opsonophagocytic assays. Samples from day 7 were used for flow cytometric analysis.
Arm/Group | 1.Aging RT | 2.Young RT | 3.Healthy Elderly | 4.Elderly DMII or HTN and Normal Renal Function | 5.Healthy Young
Number analyzed (Participants) | 9 | 10 | 12 | 9 | 8
microgram/ml
  Anti-PPS 14 IgG day 0 | 11.16 (10.52) | 9.29 (8.52) | 6.46 (5.34) | 7.69 (7.38) | 6.51 (5.6663)
  Anti-PPS14 IgG day 30 | 14.55 (10.94) | 13.92 (11.62) | 10.42 (8.04) | 13.05 (9.44) | 15.75 (10.82)
  Anti-PPS23F IgG day 0 | 3.09 (4.04) | 2.84 (3.22) | 1.10 (1.06) | 3.85 (3.73) | 2.52 (2.35)
  Anti-PPS23F IgG day 30 | 6.96 (5.39) | 4.57 (5.56) | 5.18 (3.80) | 11.55 (7.44) | 9.69 (5.11)
  Anti-PPS19A IgG day 0 | 4.79 (2.97) | 6.66 (5.79) | 5.42 (6.62) | 3.65 (5.42) | 3.42 (1.43)
  Anti-PPS 19A IgG day 30 | 14.82 (10.40) | 9.28 (6.84) | 10.43 (7.96) | 10.54 (8.83) | 8.35 (8.82)
Statistical Analysis 1: Comparison: 1.Aging RT vs 2.Young RT vs 3.Healthy Elderly vs 4.Elderly DMII or HTN and Normal Renal Function vs 5.Healthy Young; Differences between groups were compared using the paired t test; Test type: Equivalence — Differences between groups were compared using the paired t test; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: 1.Aging RT vs 2.Young RT vs 3.Healthy Elderly vs 4.Elderly DMII or HTN and Normal Renal Function vs 5.Healthy Young; Test type: Superiority; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: 1.Aging RT vs 2.Young RT vs 3.Healthy Elderly vs 4.Elderly DMII or HTN and Normal Renal Function vs 5.Healthy Young; Test type: Superiority; p < 0.05, t-test, 2 sided

2. Primary Outcome: Opsonophagocytic Antibody Titer Serum Dilution Difference Between Healthy Elderly, Elderly With DM/HTN and Elderly With RT.
Description: Measure the serum opsonophagocytic activity against streptococcus pneumonia serotypes 14, 19A and 23F on days 0 and 30 by opsonophagocytic assay.
Time Frame: Baseline and 30 days
Population: Healthy elderly versus elderly with DM versus elderly with RT
Measure: Mean (Standard Deviation); unit: titer
Groups:
- 5.Healthy Young: Healthy persons between the ages 35-45 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  13 valent conjugated pneumococcal vaccine: FDA approved pneumococcal polysaccharide vaccine containing capsular polysaccharide of 13 different pneumococcal serotypes conjugated to CRM197 was administered on day 0. Only group 5 received this as an intervention. In all other groups Prevnar 13 was given as standard of care.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples obtained from days 0 and 30 were used for antibody titers and opsonophagocytic assays. Samples from day 7 were used for flow cytometric analysis.
Arm/Group | 1.Aging RT | 2.Young RT | 3.Healthy Elderly | 4.Elderly DMII or HTN and Normal Renal Function | 5.Healthy Young
Number analyzed (Participants) | 9 | 10 | 12 | 9 | 8
titer
  opsonophagocytic titer PPS 14 day 0 | 1081 (2810) | 147 (295) | 3024 (6478) | 256 (663) | 811 (2451)
  opsonophagocytic titer PPS14 day 30 | 3117 (5860) | 275 (552) | 5954 (8117) | 2477 (4857) | 3687 (7288)
  opsonophagocytic titer PPS23F day 0 | 3.4 (2.8) | 28 (77) | 6.3 (6.3) | 3.3 (4.1) | 29 (56)
  opsonophagocytic titer PPS23F day 30 | 617 (1617) | 38 (64) | 1455 (4822) | 469 (904) | 914 (2310)
  opsonophagocytic titer PPS19A day 0 | 633 (1891) | 7 (10) | 15 (21) | 663 (2324) | 461 (1407)
  opsonophagocytic titer PPS 19A day 30 | 3893 (7711) | 138 (231) | 4529 (7549) | 4634 (7597) | 2290 (5462)
Statistical Analysis 1: Comparison: 1.Aging RT vs 2.Young RT vs 3.Healthy Elderly vs 4.Elderly DMII or HTN and Normal Renal Function vs 5.Healthy Young; Test type: Superiority; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: 1.Aging RT vs 3.Healthy Elderly vs 4.Elderly DMII or HTN and Normal Renal Function; Test type: Superiority; p < 0.05, t-test, 2 sided

3. Primary Outcome: Percentage of Polysaccharide Specific B Cells (% Cells/mL)
Description: percentage of polysaccharide specific B cells, and percentage of IgM memory B cells/mL in % cells/mL induced by vaccination with PCV13
Time Frame: day 7
Population: Participants who completed PCV13 immunization and from whom blood samples were obtained on day 0, 7, and 30.
  Elderly healthy versus elderly with DM/HTN and elderly RT
Measure: Geometric Mean (Standard Deviation); unit: percentage cells/mL
Groups:
- 1.Aging RT: Renal transplant recipients between 65-75 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause of renal failure was either DMII or HTN.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples from day 7 were used for flow cytometric analysis.
- 2.Young RT: Renal transplant recipients between 35-45 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause of renal failure was either DMII or HTN.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples from day 7 were used for flow cytometric analysis.
- 3.Healthy Elderly: Healthy persons between the ages 65-75 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23).
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples from day 7 were used for flow cytometric analysis.
- 4.Elderly DMII or HTN and Normal Renal Function: Persons between the ages 65-75 with DMII or hypertension but normal renal function who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples from day 7 were used for flow cytometric analysis.
- 5.Healthy Young: Healthy persons between the ages 35-45 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  13 valent conjugated pneumococcal vaccine: FDA approved pneumococcal polysaccharide vaccine containing capsular polysaccharide of 13 different pneumococcal serotypes conjugated to CRM197 was administered on day 0. Only group 5 received this as an intervention. In all other groups Prevnar 13 was given as standard of care.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples from day 7 were used for flow cytometric analysis.
Arm/Group | 1.Aging RT | 2.Young RT | 3.Healthy Elderly | 4.Elderly DMII or HTN and Normal Renal Function | 5.Healthy Young
Number analyzed (Participants) | 9 | 10 | 12 | 9 | 8
percentage cells/mL
  % of lymphocytes that are CD19+ (B cells) | 9.87 (5.85) | 5.31 (2.31) | 9.75 (4.05) | 7.91 (3.25) | 10.77 (4.4)
  % of CD19+ B cells that were PPS14+ post-immunization | 2.12 (0.99) | 1.55 (1.29) | 1.68 (0.75) | 1.82 (1.11) | 1.67 (0.92)
  % of CD19+ B cells that were PPS23F+ post-immunization | 1.65 (1.24) | 1.79 (1.47) | 1.22 (0.78) | 1.52 (1.01) | 1.29 (0.96)
  PPS14+ B cells that were IgM+ memory B cells day 7 post-immunization | 18.73 (16.12) | 22.95 (19.53) | 20.57 (8.49) | 24.59 (15.58) | 20.62 (10.2)
  % PPS14+ B cells that were switched memory B cells 7 d. post-immunization | 41.48 (17.31) | 51.6 (25.31) | 51.23 (17.72) | 52.46 (19.22) | 44.87 (18.33)
  %PPS23F+ B cells that were IgM memory B cells d7 post-immunization | 30.56 (12.34) | 14.67 (8.44) | 24.21 (16.66) | 32.22 (24.95) | 18.11 (10.97)
  % PPS23 F B cells that were switched memory B cells d.7 post-immunization | 40.02 (6.23) | 35.52 (14.17) | 52.48 (19.35) | 47.7 (19.71) | 49.26 (27.22)
Statistical Analysis 1: Comparison: 1.Aging RT vs 3.Healthy Elderly vs 4.Elderly DMII or HTN and Normal Renal Function; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Inflammatory Markers Serum Levels Pre-immunization
Description: Measure level of inflammatory markers BAFF, APRIL, IL6, TNF alpha and sCD40L in serum in pg/mL pre-immunization.
Time Frame: Day 0 pre-immunization
Population: Participants who completed immunization and a minimal of 30 day follow up.
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Groups:
- 1.Aging RT: Renal transplant recipients between 65-75 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause of renal failure was either DMII or HTN.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples from day 0 were used for measuring inflammatory markers.
- 2.Young RT: Renal transplant recipients between 35-45 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause of renal failure was either DMII or HTN.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples from day 0 were used for measuring inflammatory markers.
- 3.Healthy Elderly: Healthy persons between the ages 65-75 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples from day 0 were used for measuring inflammatory markers.
- 4.Elderly DMII or HTN and Normal Renal Function: Persons between the ages 65-75 with DMII or hypertension but normal renal function who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples from day 0 were used for measuring inflammatory markers.
- 5.Healthy Young: Healthy persons between the ages 35-45 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  13 valent conjugated pneumococcal vaccine: FDA approved pneumococcal polysaccharide vaccine containing capsular polysaccharide of 13 different pneumococcal serotypes conjugated to CRM197 was administered on day 0. Only group 5 received this as an intervention. In all other groups Prevnar 13 was given as standard of care.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) Samples from day 0 were used for measuring inflammatory markers.
Arm/Group | 1.Aging RT | 2.Young RT | 3.Healthy Elderly | 4.Elderly DMII or HTN and Normal Renal Function | 5.Healthy Young
Number analyzed (Participants) | 9 | 10 | 12 | 9 | 8
pg/mL
  BAFF serum concentration | 0.59 (0.10) | 0.56 (0.17) | 0.57 (0.16) | 0.58 (0.29) | 0.50 (0.08)
  APRIL serum concentration | 664.84 (206.68) | 664.84 (206.68) | 852.66 (216.65) | 870.09 (139.29) | 619.54 (161.68)
  sCD40L serum concentration | 199.25 (372.37) | 663.12 (899.98) | 984.92 (1292.38) | 1272.35 (1229.85) | 1639.47 (1356.06)
  TNFalpha serum concentration | 11.22 (7.82) | 23.96 (18.89) | 23.05 (22.52) | 20.35 (16.78) | 19.44 (16.77)
  IL6 serum concentration | 1.21 (0.83) | 2.58 (1.68) | 1.71 (1.94) | 1.21 (0.48) | 1.56 (1.64)
Statistical Analysis 1: Comparison: 1.Aging RT vs 2.Young RT vs 3.Healthy Elderly vs 4.Elderly DMII or HTN and Normal Renal Function vs 5.Healthy Young; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the duration of the duration of enrollment thus varying from participant to participant.
Description: Adverse events were collected starting at day 7, 1 month, 6 months, 1 year, varying per participant depending on duration of enrollment. Adverse events were collected from every participant enrolled, including those that dropped out of the study after their initial immunization and blood draw..
Groups:
- 1.Aging RT: Renal transplant recipients between 65-75 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause or renal failure was either DMII or HTN.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) .
- 2.Young RT: Renal transplant recipients between 35-45 years of age, on stable immunosuppression. who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23). Cause or renal failure was either DMII or HTN.
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) .
- 3.Healthy Elderly: Healthy persons between the ages 65-75 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) .
- 4.Elderly DMII or HTN and Normal Renal Function: Persons between the ages 65-75 with DMII or hypertension but normal renal function who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine (pneumovax23)
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) .
- 5.Healthy Young: Healthy persons between the ages 35-45 who previously (>1 year prior) received the 23 valent pneumococcal polysaccharide vaccine
  Peripheral blood sample: Peripheral blood samples (30-60 mL) were collected at day 0 (pre-immune), day 7, and day 30 (4 weeks post-PPV23) .
Arm/Group | 1.Aging RT | 2.Young RT | 3.Healthy Elderly | 4.Elderly DMII or HTN and Normal Renal Function | 5.Healthy Young
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12 | 0/15 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12 | 0/15 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/12 | 0/15 | 0/11 | 0/10

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of enrolled subjects due to the COVID pandemic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT03802994/Prot_SAP_000.pdf